CLINICAL TRIAL: NCT00002789
Title: A PHASE III RANDOMIZED STUDY COMPARING G-CSF MOBILIZED PERIPHERAL BLOOD STEM CELLS WITH MARROW AS THE SOURCE OF STEM CELLS FOR ALLOGENEIC TRANSPLANTS FROM HLA IDENTICAL, RELATED DONORS FOR THE TREATMENT OF CHRONIC MYELOID LEUKEMIA
Brief Title: Bone Marrow or Peripheral Stem Cell Transplantation in Treating Patients With Chronic Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 1092.00; FHCRC-1092.00; NCI-H96-0926; CDR0000064853 (Registry Identifier: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-03-19 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Leukemia
Keywords: chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; Philadelphia chromosome positive chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Busulfan; Cyclophosphamide; Cyclosporine; Methotrexate; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Drug: methotrexate
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Peripheral stem cell or bone marrow transplantation may be able to replace immune cells that were destroyed by chemotherapy used to kill tumor cells. Sometimes the transplanted cells can make an immune response against the body's normal tissues. Stem cells that have been treated in the laboratory with filgrastim may prevent this from happening. Combining chemotherapy with bone marrow or peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. It is not yet known which treatment is more effective for chronic myeloid leukemia.

PURPOSE: Randomized phase III trial to compare the effectiveness of donor peripheral stem cell transplantation with donor bone marrow transplantation in treating patients with chronic myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the incidence of persistent cytogenetic or hematologic relapse in patients with chronic myeloid leukemia in chronic or accelerated phase treated with transplantation using filgrastim (G-CSF)-mobilized peripheral blood stem cells vs bone marrow from HLA-identical, related donors. II. Compare survival and nonrelapse mortality in patients treated with these regimens. III. Compare incidence and severity of acute and chronic graft versus host disease in patients treated with these regimens. IV. Compare hospitalization and treatment associated expenses for patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age (15-39 vs 40-65), interval from diagnosis to transplantation (under 2 years vs 2 years or more, and permutations of patient and donor gender. Patients are randomized to one of two treatment arms. Arm I: Patients receive a preparative regimen comprising busulfan orally or IV 4 times daily on days -7 to -4 and cyclophosphamide IV on days -3 and -2. Allogeneic filgrastim (G-CSF)-mobilized peripheral blood stem cells are infused on day 0. Arm II: Busulfan and cyclophosphamide are administered as in arm I. Allogeneic bone marrow is infused on day 0. Patients receive graft-versus-host disease prophylaxis comprising methotrexate IV on days 1, 3, 6, and 11 and cyclosporine IV over 1-4 hours or orally every 12 hours on days -1 to 80 and then tapered. Patients are followed every 6 months for 2 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of chronic myeloid leukemia (CML) in chronic phase No chromosomal abnormalities other than a single Philadelphia chromosome (Ph) and less than 10% blasts in bone marrow and peripheral blood OR Diagnosis of CML in accelerated phase Must meet 1 of the following criteria: More than 10% and less than 30% myeloblasts plus promyelocytes in bone marrow or peripheral blood Major perturbations of WBC, platelet count, or hematocrit uncontrolled by chemotherapy with busulfan or hydroxyurea Progressive splenomegaly Extramedullary tumor Presence of any nonconstitutional cytogenetic abnormality in addition to a single Ph chromosome Persistent unexplained fever or bone pain Ph positive OR bcr/abl positive by reverse-transcriptase polymerase chain reaction or Southern blot No CML in blast phase

PATIENT CHARACTERISTICS: Age: 15 to 65 Performance status: Not specified Life expectancy: At least 6 months based on any concurrent nonmalignant disease Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2 times upper limit of normal (ULN) (unless due to CML) SGOT and SGPT no greater than 2 times ULN (unless due to CML) Renal: Creatinine no greater than 1.4 mg/dL Cardiovascular: Cardiac ejection fraction at least 45% Pulmonary: DLCO at least 50% predicted Other: HIV negative Donor Entry Criteria: HLA-identical family member No psychological, physiological, or medical condition that would preclude harvest of peripheral blood stem cells or bone marrow HIV negative Hepatitis A, B, and C antigen negative Negative pregnancy test Age 12 years and over

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 1996-05; Primary Completion 2001-09 (Actual); Study Completion 2001-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Radich, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States